CLINICAL TRIAL: NCT05977062
Title: Sleep-4-all-2.0 Study: Optimization of an Online Stepwise Therapeutic Device Based on a Cognitive-behavioral Approach for Cancer Patients With Insomnia - A Prospective Real-life Study
Brief Title: Optimization of an Online Stepwise Therapeutic Device Based on a Cognitive-behavioral Approach for Cancer Patients With Insomnia
Acronym: Sleep-4-All-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A01891-40; 2021/3317 (Other: CSET number)
Record Dates: First submitted 2023-05-24; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Cancer; Insomnia
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coaching arm (Other)
  Interventions: Other: Self screening; Other: Phone call; Other: Online questionnaires

INTERVENTIONS:
Other: Self screening — Score ISI (Index de Sévérité de l'Insomnie)
Other: Phone call — Phone call at the beginning of the program and at the middle and at the end.
Other: Online questionnaires — To be completed at week 1, 6, 12 and 24.

SUMMARY:
Determine who can benefit from additional follow-up by a professional and what type of help is most appropriate (need and expectation of patients in terms of support by a health professional)

ELIGIBILITY:
Inclusion Criteria:

* Adults patients,
* With a diagnosis of localized or metastatic cancer,
* During or after their treatment,
* In one of the following three cancer centres: Gustave Roussy (Villejuif), Montpellier Cancer Institute (Montpellier), and Léon Bérard Center (Lyon)
* With a significative score on the self-screening Insomnia Severity Index score (ISI ≥ 8)
* Able to readily read and understand French,
* Able to use informatic tools confidently and with Internet access,
* Who have signed the online consent form,
* Affiliated to a social security system or beneficiary of the same.

Exclusion Criteria:

* Patient with a visual, hearing or cognitive disability that is incompatible with the study,
* Simultaneous participation in another study evaluating a treatment of insomnia,
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-10-13 (Estimated); Study Completion 2024-10-13 (Estimated)

PRIMARY OUTCOMES:
Evolution of the ISI score | until 24 weeks after enrolment
  The primary outcome is to evaluate the evolution of the ISI score of patients with score > 8.
  ISI = Index de Sévérité de l'Insomnie. Score > 8 means the patient has insomnia issue.
Patient insomnia perception | until 24 weeks after enrolment
  Two ad-hoc items will be proposed to the participants to determine if insomnia is considered as a problem for them (outcome perception), and as a problem important to solve (outcome expectancy).
Adherence to the intervention | until 24 weeks after enrolment
  The frequency and the evolution of connections (A/globally, namely total number of connections per week and during all the intervention; B/potential differences in the frequency of connections throughout the weeks);
  * the type and proportion of components effectively consulted (videos, modules, and tools);
  * the duration of the use of the study web platform (total number of weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Diane BOINON, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (3):
- France (3):
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de Montpellier, Montpellier
  - Gustave Roussy, Villejuif